CLINICAL TRIAL: NCT03087799
Title: Brief Behavioral Treatment for Sleep Problems in Irritable Bowel Syndrome: a Pilot Study
Brief Title: Brief Behavioral Treatment for Sleep Problems in IBS Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Lembo, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000440
Record Dates: First submitted 2017-03-02; First posted 2017-03-23 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Irritable Bowel Syndrome; Sleep Disturbance
MeSH Terms: conditions — Irritable Bowel Syndrome; Parasomnias | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Behavioral Treatment for Sleep (Experimental)
  Interventions: Behavioral: Brief Behavioral Treatment for Sleep
- Wait List Control (No Intervention)

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment for Sleep — The BBT arm will consist of 2 in-person treatment visits and 2 telephone check-in visits. Treatment will involve psychoeducation about sleep hygiene and stimulus control as well as sleep schedule modification and sleep restriction. The treatment manual is attached for clarification. This manual is used solely to guide clinical decision making and will not be provided to participants.
  Arms: Brief Behavioral Treatment for Sleep

SUMMARY:
Patients with Irritable Bowel Syndrome (IBS) often report more fatigue and sleep disturbances compared to their healthy counterparts and compared to patients with other GI disorders. This pilot study will evaluate the feasibility of a Brief Behavioral Treatment for Insomnia (BBT-I) in Irritable Bowel Syndrome. 40 participants will be recruited; 20 will receive 4 weeks of BBT and 20 will be assigned to a wait list control group (WLC). The primary aim of the current project is to assess feasibility of administering BBT-I to a sample of patients with IBS. Because behavioral sleep treatment has not yet been studied in IBS or any other GI population, this project will provide information about treatment adherence, recruitment, and effect sizes. Secondary aims include evaluating the impact of BBT-I on sleep quality and IBS symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50
* Meet diagnostic criteria for IBS
* Stable medication for IBS for at least 1 month
* Stable medication for sleep for at least 1 month
* ISI cutoff score of 10 or higher
* Completes at least 5 out of 7 days of daily symptom and sleep diary during 1 week baseline

Exclusion Criteria:

* Medical history of significant head injury or other neurological disorder
* Pregnancy (self-reported)
* Post-menopause
* Major concomitant medical conditions
* Major psychiatric diagnosis with comorbid sleep problems
* Taking medications that might interfere with sleep
* Confirmed or suspected other untreated sleep disorder
* Active illicit drug use

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Change in Irritable Bowel Syndrome Severity Scoring System | 5 weeks
  A measure of IBS symptom severity

SECONDARY OUTCOMES:
Change in Insomnia Severity Index | 5 weeks
  A measure of insomnia
Change in Pittsburgh Sleep Quality Index | 5 weeks
  A measure of sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No